CLINICAL TRIAL: NCT05275153
Title: Effectiveness of a Home-Based Cognitive Rehabilitation Program Driven by a Tablet Application in Patients With Mild Cognitive Impairment
Brief Title: Effectiveness of a Home-Based Cognitive Rehabilitation Program in Patients With MCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Collaborators: Woorisoft (Unknown)
Responsible Party: Principal Investigator, Yong-il Shin, Professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02-2019-018
Record Dates: First submitted 2022-03-02; First posted 2022-03-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Cognitive Impairment; Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home based cognitive rehabilitation program (Experimental): The intervention was conducted for 30 minutes each time, 3 times a week for 8 weeks, a total of 24 times.
  Interventions: Other: Home based cognitive rehabilitation program
- No intervention (No Intervention): In the control group, natural cognitive changes with the passage of time were observed.

INTERVENTIONS:
Other: Home based cognitive rehabilitation program — The home based cognitive rehabilitation program intervention was conducted for 30 minutes each time, 3 times a week for 8 weeks, a total of 24 times.
  Arms: Home based cognitive rehabilitation program

SUMMARY:
In this study, a more specific and systematic Home-Based Cognitive Rehabilitation Program Driven by a Tablet Application is developed and the purpose of the program is to check whether cognitive function is improved when the program is applied to patients with MCI.

DETAILED DESCRIPTION:
The subjects of recruitment were the elderly with mild cognitive impairment living in the local community. Assessments were conducted 7 days before and after the intervention. Subjects received Korean-Montreal Cognitive Assessment(MoCA), semantic verbal emory test (SVLT), number memorization test; Digit Span Test (DST), category word fluency test (CWFT), phonemic word fluency test (PWFT), Korean-mini mental state test (K-MMSE), and geriatric depression scale (GDS) before and 8 weeks after the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women over the age of 55
2. Those who have visual and auditory abilities without difficulties in conducting this research
3. Those with K-MMSE (Korean-Mini Mental State Examination) score of 24 or higher and 16≤K-MoCA score<23
4. In the case of patients taking dementia treatment, those who have the same treatment regimen and dose for 3 months or more from the screening date
5. A person who can understand and respond to the questionnaire questions.
6. A person who voluntarily decided to participate in this study and gave written consent to the informed consent form

Exclusion Criteria:

1. Those with a history of alcohol or drug abuse,
2. Those with a past history of uniaxial psychiatric disorders, including intellectual disability, schizophrenia, alcoholism, and bipolar disorder
3. A person who is unable to communicate
4. Those who show all neurological symptoms that cause cognitive decline, such as Parkinson's disease, cerebral hemorrhage, brain tumor, and hydrocephalus
5. Those with a record of being unconscious for more than 1 hour due to head trauma or mild repetitive head trauma
6. Those with symptoms of depression that may affect cognitive function

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-04-22 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-08-02 (Actual)

PRIMARY OUTCOMES:
Change of the Korean-Montreal cognitive assessment(MoCA) score | Baseline and Week 8
  It is a tool to evaluate overall cognitive function. Possible scores range from 0(lowest cognitive function) to 30 (highest cognitive function). Change = Paired t-test with baseline score and week 8 score.

SECONDARY OUTCOMES:
Change of the semantic verbal emory test (SVLT) score | Baseline and Week 8
  It is a tool to evaluate language memory function. Possible scores range from 0(lowest) to 36 (highest). Change = Paired t-test with baseline score and week 8 score.
Change of the Digit Span Test (DST) score | Baseline and Week 8
  It is a tool to evaluate number memorization and attention. Possible scores range from 0(lowest) to 9 (highest). Change = Paired t-test with baseline score and week 8 score.
Change of the category word fluency test (CWFT) score | Baseline and Week 8
  It is a tool to evaluate executive function. In one minute, the speak words of the given category is performed, and the number of words spoken within the time is evaluated as a score. Change = Paired t-test with baseline score and week 8 score.
Change of the phonemic word fluency test (PWFT) score | Baseline and Week 8
  It is a tool to evaluate executive function. In one minute, the speak words that start with a given phoneme is performed, and the number of words spoken within the time is evaluated as a score. Change = Paired t-test with baseline score and week 8 score.
Change of the geriatric depression scale (GDS) score | Baseline and Week 8
  It is a tool to evaluate degree of depression. Possible scores range from 0(lowest depression) to 21 (highest depression). Change = Paired t-test with baseline score and week 8 score.

CONTACTS AND LOCATIONS:
Overall Officials: Young-Il Shin, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Pusan national university Yangsan Hospital, Gyeongsang, Yangsan, South Korea

IPD SHARING:
Plan to Share IPD: No